CLINICAL TRIAL: NCT00765011
Title: A Phase II Trial With Radiotherapy Plus Cetuximab to Evaluate Specific Survival Free of Laryngectomy in Patients With Resectable and Locally Advanced Larynx Cancer, After Treatment With TPF
Brief Title: TPF Plus Radiotherapy and Cetuximab to Avoid Total Laryngectomy in Patients With Larynx Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Tratamiento de Tumores de Cabeza y Cuello (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TTCC-2007-02
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): TPF plus concomitant treatment with cetuximab and conventional radiotherapy
  Interventions: Drug: TPF, radiotherapy and cetuximab
- Grupo B (Other): Surgery
  Interventions: Procedure: H&N surgery

INTERVENTIONS:
Drug: TPF, radiotherapy and cetuximab — 3 cycles of: cisplatin: 75mg/m2, i.v., 1 hour, once daily docetaxel: 75 mg/m2, i.v., 1 hour, once daily 5-fluorouracilo: 750 mg/m2, i.v., 24 hours, 5 days Radiotherapy: 70Gy,divided into daily doses of 2 Gray (total days:35) Cetuximab: 400 mg/m2, i.v, 2 hours, 1 day Cetuximab: 250 mg/m2, i.v, 1 hour, 7 days
  Other Names: TPF plus radiotherapy and cetuximab
  Arms: Group A
Procedure: H&N surgery — Rescue surgery
  Other Names: Rescue surgery
  Arms: Grupo B

SUMMARY:
A Phase II Trial With Radiotherapy Plus Cetuximab to Evaluate Specific Survival Free of Laryngectomy in Patients With Resectable and Locally Advanced Larynx Cancer, After Treatment With TPF Chemotherapy.

DETAILED DESCRIPTION:
This study is being sponsored by a cooperative medical group.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form.
2. Men or women, age (18 and 70).
3. ECOG scale:0-1.
4. Life expectancy superior to 3 months.
5. Larynx squamous carcinoma histologically demonstrated.
6. Patients with larynx squamous carcinoma, stage III-IVA, with resectable disease whose surgery will imply a total laryngectomy. The T should be a T3, T4A, or a T2 not candidate for a partial laryngectomy. In case of T2 of any of both locations it will be required a III or IVA stadium.
7. Patients to be able to receive treatment with TPF followed by normofractionated radiotherapy with cetuximab.
8. Measurable disease (OMS criteria).
9. Neutrophils superior or equal to 1500/mm3, platelets superior or equal to 150.000/mm3, hemoglobin superior or equal to 10 g/dl.
10. Adequate renal function: creatinin lower or equal to 120 µmol/l (1,4mg/dl)
11. Adequate hepatic function: bilirubin lower or equal to 1 x UNL, AST and ALT lower or equal to 2,5 UNL, alkaline phosphatase lower or equal to 5 UNL.
12. Seric calcium adjusted to albumine lower or equal to 1,25 UNL.
13. Adequate nutritional condition: loss of weight <20% with relation to the theoretical weight and albumin superior or equal to 35 g/L.
14. Use of an effective contraceptive method.

Exclusion Criteria:

1. Metastatic disease
2. Surgical treatment, previous radiotherapy and/or chemotherapy for the study disease.
3. Other tumour locations in H&N that are not larynx.
4. Other stages that are not III or IVa without metastasis and resectable disease.
5. The following cases, which will be considered candidates for radical surgery, will not be included in the study:

   * Tumors of the subglottis.
   * Tumors of glottis or supraglottis with subglottal extension
   * Tumor that destroys the thyroid cartilage and/or cricoid and it extends to thyroid gland or soft necks's tissues.
   * Tumor of supraglottis with a superior extension to 1 cm towards the tongue base (the extension will be measured since the vallecula).
6. Other previous and/or synchronic squamous carcinoma.
7. Diagnosis of another neoplasia in the last 5 years, excepting carcinoma in situ of uterine neck and/or a cutaneous carcinoma basocellular properly treated.
8. Active infection(at needs endovenous antibiotics), including active tuberculosis and diagnosed HIV.
9. Not controlled hypertension defined as arterial systolic tension superior or equal to 180 mm Hg and/or diastolic arterial tension superior or equal to 130 mm Hg baseline.
10. Pregnancy or breastfeeding.
11. Immunity systemic treatment, chronic and concomitant, or hormonal treatment of the cancer.
12. Other antineoplasic concomitant treatments.
13. Coronary clinically significant arteriopathy or precedents of myocardial infarction in the last 12 months or high risk of not controlled arrhythmia or cardiac not controlled insufficiency.
14. Pulmonary obstructive chronic disease that had needed 3 or more hospitalizations in the last 12 months.
15. Active non controlled peptic ulcer.
16. Presence of a psychological or medical disease that could prevent to accomplish the study by the patient or to grant his/her signature in the informed consent form.
17. Known drugs abuse (excepting excessive consumption of alcohol).
18. Known allergic reaction to some of the components of the treatment of the study.
19. Previous treatment with monoclonal antibodies or other transduction of the sign inhibitors or treatment directed against the EGFR.
20. Any experimental treatment in 30 days before entry in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2008-10; Primary Completion 2014-02 (Actual); Study Completion 2015-05-12 (Actual)

PRIMARY OUTCOMES:
Specific survival free of total laryngectomy | Three years after the end of treatment with radiotherapy and cetuximab
  Time from the start of TPF treatment to death caused by the disease or by the treatment of the disease, or even to surgery involving total laryngectomy. Deaths caused by other reasons were considered "censored" data on the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Mesía Nin, MD, Principal Investigator — Hospital Durán i Reynals; José A. García Sáenz, MD, Principal Investigator — Hospital San Carlos, Madrid
Locations (17):
- Spain (17):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Manresa, Manresa, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Dr.Josep Trueta (ICO Girona), Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Oncogranada, Granada
  - Hospital Xeral Calde, Lugo
  - Hospital Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario San Carlos, Madrid
  - Hospital Son Llátzer, Palma de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario la Fe de Valencia, Valencia
  - Hospital Clínico Universitario de Zaragoza, Zaragoza
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- See also: This site would like to expose the activities of the group and at the same time serve as an information and communication tool of this pathology for professionals and patients. — http://www.ttccgrupo.org